CLINICAL TRIAL: NCT04189796
Title: Effect of Jarlsberg Cheese Compared to Cheese Without Vitamin K2 Regarding Increased Osteocalcin Level in Healthy Women
Brief Title: Jarlsberg Cheese Compared to Camembert Cheese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Stig Larsen (Other)
Collaborators: Norwegian University of Life Sciences (Other); Tine (Industry)
Responsible Party: Sponsor-Investigator, Prof Stig Larsen, Professor, Meddoc
Organization: Meddoc (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HV-Jarlsberg/III
Record Dates: First submitted 2019-12-02; First posted 2019-12-06 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Healthy Women; Osteocalcin
Keywords: Cheese intake; Vitamin K
MeSH Terms: interventions — Cheese

STUDY DESIGN:
Intervention Model Description: The study will be performed as a randomized Norwegian multicenter study with a semi-cross over design in which the participants randomized to Camembert cheese will be switched to Jarlsberg cheese after 6 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jarlsberg (Active Comparator): Daily intake of Jarlsberg Cheese in at least 6 weeks
  Interventions: Dietary Supplement: Cheese
- Camembert (Sham Comparator): Daily intake of Camembert Cheese in 6 weeks
  Interventions: Dietary Supplement: Cheese

INTERVENTIONS:
Dietary Supplement: Cheese — Daily oral intake of cheese

SUMMARY:
The study objective consists of the following three aims:

1. To compare the effect of daily intake of Jarlsberg cheese and Camembert cheese in change of the Osteocalcin level in healthy women after 6 weeks.
2. To estimate the long-term increase of the osteocalcin level, change in the lipid pattern and the vital signs caused by optimized daily intake of Jarlsberg cheese.
3. To verify the estimated maintaining dose of Jarlsberg cheese related to stabilized osteocalcin Level.

The study population consists of Healthy Voluntary (HV) women between 20 years and pre-menopausal age. The trial will be performed as a randomized Norwegian multicenter study with a semi-cross over design in which the participants randomized to Camembert cheese will be switched to Jarlsberg cheese after 6 weeks.

DETAILED DESCRIPTION:
The recruited HV women fulfilled the inclusion without the exclusion criteria for the study will undergo a screening clinical investigation. The participants will be asked to avoid use of other cheese than the one allocated to in the study, but eat as usual. One week later, the first clinical investigation in the study will take place including blood sampling and measurement of vital signs. The HV women verified to fulfil the criteria for participation and signed the informed consent form will be included in the study. During this first clinical investigation in the study denoted as Day 0, the participants receive a study identification number. The HV will randomly be allocated to either daily intake of Jarlsberg cheese or Camembert cheese. The daily intake of cheese will be 57g/day in both study groups.

The participants meet for new clinical investigations every third week with measurement of vital signs and blood sampling. Osteocalcin and vitamin K will be analysed every third week whereas the haematological and biochemical analysis will be performed every six week.

The HVs allocated to Camembert cheese will after 6 weeks be switched to daily intake of Jarlsberg cheese in additional 6 weeks with clinical investigations every third week. The participants performed the 6 weeks of daily intake of Jarlsberg cheese will either be offered participation in the cheese de-escalation study (HV-Jarlsberg/IB) or an extended study of 6 weeks with unchanged Jarlsberg cheese dose. HVs with an increase <10% in the osteocalcin level from screening to 6 weeks of Jarlsberg cheese intake will not be offered included in the de-escalation study. The first 12 HVs finalized 6 weeks with daily intake of Jarlsberg cheese obtaining an increase in the osteocalcin level from baseline ≥10% will be allocated to the de-escalation study HV-Jarlsberg/IB (separate protocol). The HVs included in the extended part of this study will receive an unchanged daily dose of Jarlsberg cheese for additional 6 weeks with clinical investigation every third week. The HVs switched to Jarlsberg cheese may be offered participation in a study part aiming to verify the maintaining dose obtained in HV-Jarlsberg/IB study. The duration of this part will be 6 weeks with clinical investigation every third week.

The main variable in this study will be osteocalcin measured in blood serum. Additionally, carboxylated and under carboxylated Osteocalcin and the ratio OR = [Carboxylated / Under Carboxylated] osteocalcin in serum will be central together the K2 variants MK-7, 8, 9, 9(4H) and vitamin K1. Triglyceride, LDL- and HDL cholesterol, vitamin D and vital signs will be secondary variables. As safety variables, haematological- and biochemical variables and adverse events (AE) will be recorded at each visit.Totally 64 HVs completing the study will be recruited from the eight participating General Practitioners sites.

ELIGIBILITY:
Inclusion Criteria:

* heathy women from 20 years and within pre-menopausal age

Exclusion Criteria:

* Pregnant women
* Known gastrointestinal disorder
* Abnormal liver or kidney function.
* Diabetes
* Suffering from verified cancer
* Under systemic treatment with corticosteroids or other immunosuppressive drugs the last 3 weeks before start of the trial treatment.
* Participating in another clinical trial with pharmaceuticals the last six weeks before start of this trial treatment.
* Lactose intolerance or known milk product allergy
* Not able to understand information.
* Do not want or not able to give written consent to participate in the study.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Osteocalcin | 6 weeks
  measured as ng/ml in serum
Vitamin K | 6 weeks
  measured as ng/ml in serum

SECONDARY OUTCOMES:
Lipids | 6 weeks
  Total cholesterol, HDL- and LDL-cholesterol measured as mmol/L in serum
Vital signs | Every 6 weeks
  Systolic- and Diastolic bloodpressure measured in mmHg after 5 minutes in supine position

CONTACTS AND LOCATIONS:
Overall Officials: Helge E Lundberg, MD, Principal Investigator — Skjetten Medical Center
Locations (1):
- Skjetten Legesenter, Skjetten, Skedsmo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lundberg HE, Glaso M, Chhura R, Shukla AA, Austlid T, Sarwar Z, Hovland K, Iqbal S, Fagertun HE, Holo H, Larsen SE. Effect on bone anabolic markers of daily cheese intake with and without vitamin K2: a randomised clinical trial. BMJ Nutr Prev Health. 2022 Aug 2;5(2):182-190. doi: 10.1136/bmjnph-2022-000424. eCollection 2022 Dec. PMID 36619332